CLINICAL TRIAL: NCT05439096
Title: Comparative Effects of Functional Exercise Versus High Frequency Transcutaneous Electrical Nerve Stimulation on Pain and Sleep Quality in Students With Primary Dysmenorrhea
Brief Title: Effects of Functional Exercise Versus High Frequency Transcutaneous Electrical Nerve Stimulation on Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-FSD-00250
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Primary Dysmenorrhea
Keywords: Functional Exercise; High Frequency; Transcutaneous Electrical Nerve Stimulation; Primary Dysmenorrhea; Menstrual Pain; Randomized Control Trial
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Exercise (Experimental): * 2 stretching exercises
  * 1 yoga exercises
  * 2 core strengthening exercises
  * 2 pelvic area exercises
  * Kegel exercises
  * Warm up for 5 minutes the apply perform exercise 3 times a week for 8 weeks and 45 minutes duration at a time
  Interventions: Other: Functional Exercise
- High Frequency Transcutaneous Electrical Nerve Stimulation (Experimental): High frequency TENS by below mentioned parameters will be applied.
  * Pulse waveform = Biphasic waveform
  * Pulse recurrence = 50 to 120 Hz
  * Phase duration = 100 µsec
  * Current amplitudes = highest tolerable intensity with continuous adjustment
  * Skin arrangement = flawless skin region.
  * Type of electrodes = Self-adhesive
  * Size and location of electrodes = It will be adjusted specifically to each woman according to the typical area of her pain.
  Interventions: Other: High Frequency Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Functional Exercise — Among Functional Exercises, cobra position is most effective in reducing pelvic pain while others are cat and fish position.Kegel exercises along with other strengthening activities for pelvic floor muscles have been accounted for in writing to favorably affect primary dysmenorrheal.
  Arms: Functional Exercise
Other: High Frequency Transcutaneous Electrical Nerve Stimulation — Transcutaneous electrical nerve stimulation, best treat primary dysmenorrhea. Transcutaneous Electrical Nerve Stimulation is proposed as an incredible spasm decrease, lessening torment, decline of analgesics and improving personal satisfaction in primary dysmenorrhea patients.
  Arms: High Frequency Transcutaneous Electrical Nerve Stimulation

SUMMARY:
The objective of this study is to assess the impacts of utilitarian exercise versus high frequency anscutaneous Electrical Nerve Stimulation on pain and sleep quality in students with primary dysmenorrhea.

DETAILED DESCRIPTION:
A Randomized Control Trial study will be directed at Riphah International University Faisalabad after synopsis approval. The Purposive examining method will be utilized to enlist the patients. Patients will be enrolled according to the pre-characterized criteria. Sample size for this examination is 40 females (18 yrs - 30 yrs) as per determination measures. The patients of one group will recieve exercise therapy and patients of other group will recieve high frequency Transcutaneous Electrical Nerve Stimulation. The patient's result will be assessed following a month of treatment . Informed consent will be taken from each patient. Data entry and analysis will be done with Statistical Package of Social Sciences version 20.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed instance of primary dysmenorrhea
2. Age somewhere in the range of 18 and 30 years,
3. A history of lower stomach torment for in excess of 6 periods.
4. Moderate or serious torment, with a numeric rating scale (NRS) score ≥5 out of 10.
5. No elective treatment including TENS inside multi month before enlistment in the investigation; and
6. Provision of educated agree preceding enlistment in the examination.

Exclusion Criteria:

1. Pregnant or Breastfeeding,
2. History of medical procedure of the lower midsection,
3. Heart sickness,
4. Cancer,
5. Severe mental problems.
6. Those who couldn't utilize TENS, for instance, in view of a lasting pacemaker or skin infection.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females Experiencing Primary Dysmenorrhea
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12th Week
  A Visual Analogue Scale is a measurement instrument, Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No